CLINICAL TRIAL: NCT01620073
Title: Home-Based Versus Partner-Friendly Clinic Testing to Enhance Male Partner HIV-1 Testing During Pregnancy: A Randomized Clinical Trial
Brief Title: Home-Based Versus Partner-Friendly Clinic Testing to Enhance Male Partner HIV-1 Testing During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Alfred Osoti MBChB MMed, Doctor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 42561
Record Dates: First submitted 2012-06-12; First posted 2012-06-15 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Male Partner; HIV Counseling and Testing; Home Based; Pregnancy
Keywords: Male partner; HIV counseling and testing; Home based; Pregnancy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Partner friendly arm (Other): Proportion of males counseled and tested using routine standards of prenatal care
  Interventions: Other: HIV counseling and testing
- Home based arm (Experimental): Proportion of male partners accepting HIV counseling and testing following home visits for couple HIV counseling and testing during pregnancy
  Interventions: Other: HIV counseling and testing

INTERVENTIONS:
Other: HIV counseling and testing — Male partner HIV counseling and testing

SUMMARY:
The investigators hypothesize that home based HIV counseling and testing can increase male partner uptake of HIV testing during pregnancy.

The investigators study aims through a randomized clinical trial to determine whether a home-based model (HBM) versus a partner-friendly clinic model (PFM) can increase male uptake of HIV counseling and testing during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women and their male partners

Exclusion Criteria:

* Non-pregnant, minors, inability to live in study area for 6 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of Male Partners Counseled and Tested for HIV During Pregnancy | 6 weeks
  To determine male partner acceptability of counseling and testing within a six week period following the counseling and testing of the pregnant woman.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred O Osoti, MBChB MMed, Principal Investigator — University of Washington
Locations (2):
- Kenya (2):
  - Ahero Sub-District Hospital, Nyando, Kenya, Kisumu, Nyanza
  - Ahero Sub-District Hospital, Kisumu, Nyanza

REFERENCES:
- [Derived] Osoti AO, John-Stewart G, Kiarie JN, Barbra R, Kinuthia J, Krakowiak D, Farquhar C. Home-based HIV testing for men preferred over clinic-based testing by pregnant women and their male partners, a nested cross-sectional study. BMC Infect Dis. 2015 Jul 30;15:298. doi: 10.1186/s12879-015-1053-2. PMID 26223540
- [Derived] Osoti AO, John-Stewart G, Kiarie J, Richardson B, Kinuthia J, Krakowiak D, Farquhar C. Home visits during pregnancy enhance male partner HIV counselling and testing in Kenya: a randomized clinical trial. AIDS. 2014 Jan 2;28(1):95-103. doi: 10.1097/QAD.0000000000000023. PMID 23942059